CLINICAL TRIAL: NCT01420237
Title: Restoration® Anatomic Dual Mobility (ADM) X3® Acetabular System Study With Long Term Data Collection for the Accolade® II Hip Stem
Brief Title: Restoration® Anatomic Dual Mobility (ADM) X3® Acetabular System Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As longitudinal patient follow-up continues to lag, it has been determined that the study is no longer able to meet its objectives.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70
Record Dates: First submitted 2011-03-18; First posted 2011-08-19 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Noninflammatory joint disease of the hip.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restoration ADM X3 Device (Other): Restoration ADM X3 Device in total hip replacement.
  Interventions: Device: Restoration ADM X3 Device

INTERVENTIONS:
Device: Restoration ADM X3 Device — Restoration ADM X3 Device in total hip replacement.

SUMMARY:
The purpose of this study is to evaluate the success rate of cementless primary hip replacement with the Restoration® ADM X3® Acetabular System as compared to other primary hip systems in the literature, through absence of femoral head dislocation at 10 years postoperative.

DETAILED DESCRIPTION:
This study is a prospective, open-label, post-market, non-randomized, multi-center, clinical evaluation of the Restoration® ADM X3® Acetabular System for primary total hip arthroplasty (THA) with a cementless application in a consecutive series of patients who meet the eligibility criteria. The total enrollment goal for the study is 350 cases, all of which will receive the Restoration® ADM X3® Acetabular System. A minimum of 100 cases (within the study population) will receive the Accolade® II Hip Stem. The remaining cases will receive any other compatible Stryker femoral component.

Data in the literature from other primary hip systems and similar dual mobility cups will be used as historical references.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an IRB/EC approved, study specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female, skeletally mature and age 18-75 years at time of study device implantation.
* Patient has a diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
* Patient is a candidate for a primary cementless acetabular replacement.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) ≥ 40.
* Patient has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* Patient requires revision surgery of a previously implanted total hip replacement or hip fusion to the affected joint.
* Patient has a known sensitivity to device materials.
* Patient is a prisoner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2011-06; Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hedley, M.D., Principal Investigator — Arizona Institute for Bone & Joint Disorders; Kipling Sharpe, M.D., Principal Investigator — OrthoArizona; Craig J. Della Valle, M.D., Principal Investigator — Rush University Medical Center; Geoffrey Westrich, M.D., Principal Investigator — Hospital for Special Surgery, New York; Joseph Nessler, M.D., Principal Investigator — St. Cloud Orthopedic Associates; Brian C de Beaubien, M.D., Principal Investigator — Covenant Medical Center; Christoph Lohmann, MD, Principal Investigator — Universitatsklinikum Madgeburg A.o.R.; Paul Kim, MD, Principal Investigator — The Ottawa Hospital; Amit Atrey, MD, Principal Investigator — Unity Health Toronto; Brett Greenky, MD, Principal Investigator — Syracuse Orthopedic Specialists; Ajay Aggarwal, MD, Principal Investigator — Missouri Orthopaedic Institute; Edward Petrow, DO, Principal Investigator — Tucson Orthopaedic Institute
Locations (12):
- United States (9):
  - OrthoArizona, Gilbert, Arizona
  - Arizona Institute for Bone and Joint Disorders, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Rush University Medical Center, Chicago, Illinois
  - Covenant Medical Center, Saginaw, Michigan
  - St. Cloud Orthopedic Associates, Sartell, Minnesota
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Syracuse Orthopedic Specialists, Fayetteville, New York
  - Hospital for Special Surgery, New York, New York
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Universitatsklinikum Madgeburg A.o.R. Orthopadische Universitatsklinikum Haus 8, Magdeburg, Saxony-Anhalt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 390 hips in 367 participants that were enrolled in the study. (23 bilateral cases).
Pre-assignment Details: Of the 390 hips/367 participants enrolled there were 36 hips/34 participants censored due to not having the study device, surgery canceled or an inclusion exclusion violation so 354 hips/333 participants are followed who did receive the study device and met protocol criteria. Those applicable data are reflected in this record.
Units Other Than Participants: Hips
Period: Overall Study
Arm/Group | Restoration ADM X3 Device
Started | 367; 390 Hips
Met Protocol Inclusion Criteria | 333; 354 Hips
Completed | 67; 70 Hips
Not Completed | 300; 320 Hips
Not completed — Death | 13
Not completed — Withdrawal by Subject | 41
Not completed — Lost to Follow-up | 32
Not completed — Adverse Event | 10
Not completed — Investigative Site Termination | 43
Not completed — Censored because study device not implanted | 21
Not completed — Censored because surgery not performed | 2
Not completed — Censored because of Inclusion Exclusion Violation | 11
Not completed — Sponsor terminated study early | 127

BASELINE CHARACTERISTICS:
Population: The analysis population includes 333 participants and 354 hips.
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Age, Continuous [Mean (Full Range); unit: years] — For bilateral total hip replacement participants, the age at the time of initial hip replacement surgery is used.
  years
    Mean age | 60.99 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 315
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Defined as absence of postoperative femoral head dislocation.
Time Frame: 10 years postoperative
Population: Participants/hips with available data up to 10 years or at the time of early study termination.
Measure: Number; unit: hips
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
hips | 354

2. Secondary Outcome: Harris Hip Score (HHS) Score Improvement From Preoperative Score
Description: The Harris Hip Score (HHS) assesses pain, function, joint deformity and range of motion. Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor
Time Frame: pre-op, 6 week, 1,2,3,4,5 years. 7 and 10 years were optional.
Population: Participants/hips with available data. In addition to the outcome measure time frame detailed above, data is presented at 7 and 10 years, but these visits were optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
score on a scale
  Preoperative: number analyzed (Participants) | 327
  Preoperative: number analyzed (hips) | 346
  Preoperative | 54.47 (12.85)
  6 weeks: number analyzed (Participants) | 308
  6 weeks: number analyzed (hips) | 324
  6 weeks | 79.56 (14.03)
  1 year: number analyzed (Participants) | 274
  1 year: number analyzed (hips) | 293
  1 year | 92.32 (10.44)
  2 years: number analyzed (Participants) | 246
  2 years: number analyzed (hips) | 264
  2 years | 92.99 (10.35)
  3 years: number analyzed (Participants) | 179
  3 years: number analyzed (hips) | 193
  3 years | 94.80 (9.00)
  4 years: number analyzed (Participants) | 142
  4 years: number analyzed (hips) | 153
  4 years | 94.22 (9.06)
  5 years: number analyzed (Participants) | 157
  5 years: number analyzed (hips) | 170
  5 years | 95.66 (6.69)
  7 years: number analyzed (Participants) | 70
  7 years: number analyzed (hips) | 75
  7 years | 93.77 (9.22)
  10 years: number analyzed (Participants) | 30
  10 years: number analyzed (hips) | 30
  10 years | 95.43 (7.67)

3. Secondary Outcome: All Cause Revision and Removal Rates of the Restoration ADM X3 Acetabular System
Description: Revision or removal of any study component.
Time Frame: 10 years
Population: Includes all participants who received the study device and were not censored from analysis.
Measure: Number; unit: hips
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
hips | 12

4. Secondary Outcome: Patient Satisfaction and Pain: Follow-up Questionnaire
Description: This questionnaire will be used to obtain the following information:
  * Satisfaction with the hip replacement
  * Presence of any pain in the study hip
  * Surgeries performed on the study hip
  * Any dislocations in the study hip
Time Frame: 6-10 years
Population: Participants/hips with available data at the 6,7,8.9.10 years postoperative.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
hips
  Presence of any pain in the study hip at 6 years - Yes: number analyzed (Participants) | 187
  Presence of any pain in the study hip at 6 years - Yes: number analyzed (hips) | 197
  Presence of any pain in the study hip at 6 years - Yes | 25
  Presence of any pain in the study hip at 6 years - No: number analyzed (Participants) | 187
  Presence of any pain in the study hip at 6 years - No: number analyzed (hips) | 197
  Presence of any pain in the study hip at 6 years - No | 172
  Satisfaction with the hip replacement at 6 years - Yes: number analyzed (Participants) | 183
  Satisfaction with the hip replacement at 6 years - Yes: number analyzed (hips) | 195
  Satisfaction with the hip replacement at 6 years - Yes | 191
  Satisfaction with the hip replacement at 6 years - No: number analyzed (Participants) | 183
  Satisfaction with the hip replacement at 6 years - No: number analyzed (hips) | 195
  Satisfaction with the hip replacement at 6 years - No | 4
  Surgeries performed on the study hip at 6 years - Yes: number analyzed (Participants) | 185
  Surgeries performed on the study hip at 6 years - Yes: number analyzed (hips) | 197
  Surgeries performed on the study hip at 6 years - Yes | 0
  Surgeries performed on the study hip at 6 years - No: number analyzed (Participants) | 185
  Surgeries performed on the study hip at 6 years - No: number analyzed (hips) | 197
  Surgeries performed on the study hip at 6 years - No | 197
  Any dislocations in the study hip at 6 years - Yes: number analyzed (Participants) | 185
  Any dislocations in the study hip at 6 years - Yes: number analyzed (hips) | 197
  Any dislocations in the study hip at 6 years - Yes | 0
  Any dislocations in the study hip at 6 years - No: number analyzed (Participants) | 185
  Any dislocations in the study hip at 6 years - No: number analyzed (hips) | 197
  Any dislocations in the study hip at 6 years - No | 197
  Presence of any pain in the study hip at 7 years - Yes: number analyzed (Participants) | 154
  Presence of any pain in the study hip at 7 years - Yes: number analyzed (hips) | 163
  Presence of any pain in the study hip at 7 years - Yes | 22
  Presence of any pain in the study hip at 7 years - No: number analyzed (Participants) | 154
  Presence of any pain in the study hip at 7 years - No: number analyzed (hips) | 163
  Presence of any pain in the study hip at 7 years - No | 141
  Satisfaction with the hip replacement at 7 years - Yes: number analyzed (Participants) | 153
  Satisfaction with the hip replacement at 7 years - Yes: number analyzed (hips) | 163
  Satisfaction with the hip replacement at 7 years - Yes | 162
  Satisfaction with the hip replacement at 7 years - No: number analyzed (Participants) | 153
  Satisfaction with the hip replacement at 7 years - No: number analyzed (hips) | 163
  Satisfaction with the hip replacement at 7 years - No | 1
  Surgeries performed on the study hip at 7 years - Yes: number analyzed (Participants) | 153
  Surgeries performed on the study hip at 7 years - Yes: number analyzed (hips) | 163
  Surgeries performed on the study hip at 7 years - Yes | 0
  Surgeries performed on the study hip at 7 years - No: number analyzed (Participants) | 153
  Surgeries performed on the study hip at 7 years - No: number analyzed (hips) | 163
  Surgeries performed on the study hip at 7 years - No | 163
  Any dislocations in the study hip at 7 years - Yes: number analyzed (Participants) | 153
  Any dislocations in the study hip at 7 years - Yes: number analyzed (hips) | 163
  Any dislocations in the study hip at 7 years - Yes | 0
  Any dislocations in the study hip at 7 years - No: number analyzed (Participants) | 153
  Any dislocations in the study hip at 7 years - No: number analyzed (hips) | 163
  Any dislocations in the study hip at 7 years - No | 163
  Presence of any pain in the study hip at 8 years - Yes: number analyzed (Participants) | 120
  Presence of any pain in the study hip at 8 years - Yes: number analyzed (hips) | 129
  Presence of any pain in the study hip at 8 years - Yes | 12
  Presence of any pain in the study hip at 8 years - No: number analyzed (Participants) | 120
  Presence of any pain in the study hip at 8 years - No: number analyzed (hips) | 129
  Presence of any pain in the study hip at 8 years - No | 117
  Satisfaction with the hip replacement at 8 years - Yes: number analyzed (Participants) | 119
  Satisfaction with the hip replacement at 8 years - Yes: number analyzed (hips) | 129
  Satisfaction with the hip replacement at 8 years - Yes | 128
  Satisfaction with the hip replacement at 8 years - No: number analyzed (Participants) | 119
  Satisfaction with the hip replacement at 8 years - No: number analyzed (hips) | 129
  Satisfaction with the hip replacement at 8 years - No | 1
  Surgeries performed on the study hip at 8 years - Yes: number analyzed (Participants) | 119
  Surgeries performed on the study hip at 8 years - Yes: number analyzed (hips) | 129
  Surgeries performed on the study hip at 8 years - Yes | 0
  Surgeries performed on the study hip at 8 years - No: number analyzed (Participants) | 119
  Surgeries performed on the study hip at 8 years - No: number analyzed (hips) | 129
  Surgeries performed on the study hip at 8 years - No | 129
  Any dislocations in the study hip at 8 years - Yes: number analyzed (Participants) | 119
  Any dislocations in the study hip at 8 years - Yes: number analyzed (hips) | 129
  Any dislocations in the study hip at 8 years - Yes | 0
  Any dislocations in the study hip at 8 years - No: number analyzed (Participants) | 119
  Any dislocations in the study hip at 8 years - No: number analyzed (hips) | 129
  Any dislocations in the study hip at 8 years - No | 129
  Presence of any pain in the study hip at 9 years - Yes: number analyzed (Participants) | 77
  Presence of any pain in the study hip at 9 years - Yes: number analyzed (hips) | 81
  Presence of any pain in the study hip at 9 years - Yes | 8
  Presence of any pain in the study hip at 9 years - No: number analyzed (Participants) | 77
  Presence of any pain in the study hip at 9 years - No: number analyzed (hips) | 81
  Presence of any pain in the study hip at 9 years - No | 73
  Satisfaction with the hip replacement at 9 years - Yes: number analyzed (Participants) | 74
  Satisfaction with the hip replacement at 9 years - Yes: number analyzed (hips) | 80
  Satisfaction with the hip replacement at 9 years - Yes | 79
  Satisfaction with the hip replacement at 9 years - No: number analyzed (Participants) | 74
  Satisfaction with the hip replacement at 9 years - No: number analyzed (hips) | 80
  Satisfaction with the hip replacement at 9 years - No | 1
  Surgeries performed on the study hip at 9 years - Yes: number analyzed (Participants) | 74
  Surgeries performed on the study hip at 9 years - Yes: number analyzed (hips) | 80
  Surgeries performed on the study hip at 9 years - Yes | 0
  Surgeries performed on the study hip at 9 years - No: number analyzed (Participants) | 74
  Surgeries performed on the study hip at 9 years - No: number analyzed (hips) | 80
  Surgeries performed on the study hip at 9 years - No | 80
  Any dislocations in the study hip at 9 years - Yes: number analyzed (Participants) | 74
  Any dislocations in the study hip at 9 years - Yes: number analyzed (hips) | 80
  Any dislocations in the study hip at 9 years - Yes | 0
  Any dislocations in the study hip at 9 years - No: number analyzed (Participants) | 74
  Any dislocations in the study hip at 9 years - No: number analyzed (hips) | 80
  Any dislocations in the study hip at 9 years - No | 80
  Presence of any pain in the study hip at 10 years - Yes: number analyzed (Participants) | 67
  Presence of any pain in the study hip at 10 years - Yes: number analyzed (hips) | 70
  Presence of any pain in the study hip at 10 years - Yes | 8
  Presence of any pain in the study hip at 10 years - No: number analyzed (Participants) | 67
  Presence of any pain in the study hip at 10 years - No: number analyzed (hips) | 70
  Presence of any pain in the study hip at 10 years - No | 62
  Satisfaction with the hip replacement at 10 years - Yes: number analyzed (Participants) | 67
  Satisfaction with the hip replacement at 10 years - Yes: number analyzed (hips) | 70
  Satisfaction with the hip replacement at 10 years - Yes | 69
  Satisfaction with the hip replacement at 10 years - No: number analyzed (Participants) | 67
  Satisfaction with the hip replacement at 10 years - No: number analyzed (hips) | 70
  Satisfaction with the hip replacement at 10 years - No | 1
  Surgeries performed on the study hip at 10 years - Yes: number analyzed (Participants) | 67
  Surgeries performed on the study hip at 10 years - Yes: number analyzed (hips) | 70
  Surgeries performed on the study hip at 10 years - Yes | 1
  Surgeries performed on the study hip at 10 years - No: number analyzed (Participants) | 67
  Surgeries performed on the study hip at 10 years - No: number analyzed (hips) | 70
  Surgeries performed on the study hip at 10 years - No | 69
  Any dislocations in the study hip at 10 years - Yes: number analyzed (Participants) | 67
  Any dislocations in the study hip at 10 years - Yes: number analyzed (hips) | 70
  Any dislocations in the study hip at 10 years - Yes | 0
  Any dislocations in the study hip at 10 years - No: number analyzed (Participants) | 67
  Any dislocations in the study hip at 10 years - No: number analyzed (hips) | 70
  Any dislocations in the study hip at 10 years - No | 70

5. Secondary Outcome: Radiographic Stability Rates
Description: Cases that present with migration of greater than 5 mm in any direction or at least 2 mm radiolucency in all zones will be considered radiographic failures. All cases were assessed for any migration at the 6 week, 1,2,3,4,5 year time points.
Time Frame: 6 week,1, 2, 3, 4, 5 years
Population: Participants/hips with available radiographic data submitted at the outcome measure time frames.
Measure: Number; unit: hips
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
hips | 0

6. Secondary Outcome: Complication Rates for Psoas Impingement and Associated Groin Pain
Description: Reported occurrence of any participant/hip experiencing groin pain or psoas impingement.
Time Frame: 10 years
Population: Participants/hips that reported an event of groin pain or psoas impingement up until early study termination.
Measure: Number; unit: hips
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
hips | 2

7. Secondary Outcome: Short Form-12 (SF-12) Improvement From Preoperative Score
Description: The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: preop, 6 week, 1,2,3,4,5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
score on a scale
  Pre-op Physical Component | 32.62 (8.94)
  6 weeks Physical Component: number analyzed (Participants) | 315
  6 weeks Physical Component: number analyzed (hips) | 333
  6 weeks Physical Component | 40.02 (8.49)
  1-year Physical Component: number analyzed (Participants) | 286
  1-year Physical Component: number analyzed (hips) | 306
  1-year Physical Component | 48.43 (9.6)
  2-years Physical Component: number analyzed (Participants) | 257
  2-years Physical Component: number analyzed (hips) | 276
  2-years Physical Component | 49.44 (8.63)
  3-years Physical Component: number analyzed (Participants) | 221
  3-years Physical Component: number analyzed (hips) | 238
  3-years Physical Component | 49.69 (8.79)
  4-years Physical Component: number analyzed (Participants) | 201
  4-years Physical Component: number analyzed (hips) | 217
  4-years Physical Component | 48.93 (9.31)
  5-years Physical Component: number analyzed (Participants) | 200
  5-years Physical Component: number analyzed (hips) | 214
  5-years Physical Component | 48.49 (9.73)
  7-years Physical Component: number analyzed (Participants) | 121
  7-years Physical Component: number analyzed (hips) | 130
  7-years Physical Component | 48.45 (9.39)
  10-years Physical Component: number analyzed (Participants) | 51
  10-years Physical Component: number analyzed (hips) | 54
  10-years Physical Component | 49.26 (8.86)
  Pre-op Mental Component | 52.42 (10.99)
  6 weeks Mental Component: number analyzed (Participants) | 315
  6 weeks Mental Component: number analyzed (hips) | 333
  6 weeks Mental Component | 55.18 (9.33)
  1-year Mental Component: number analyzed (Participants) | 286
  1-year Mental Component: number analyzed (hips) | 306
  1-year Mental Component | 55.2 (7.61)
  2-years Mental Component: number analyzed (Participants) | 257
  2-years Mental Component: number analyzed (hips) | 276
  2-years Mental Component | 54.88 (7.8)
  3-years Mental Component: number analyzed (Participants) | 221
  3-years Mental Component: number analyzed (hips) | 238
  3-years Mental Component | 54.92 (7.69)
  4-years Mental Component: number analyzed (Participants) | 201
  4-years Mental Component: number analyzed (hips) | 217
  4-years Mental Component | 55.85 (6.95)
  5-years Mental Component: number analyzed (Participants) | 200
  5-years Mental Component: number analyzed (hips) | 214
  5-years Mental Component | 55.29 (7.81)
  7-years Mental Component: number analyzed (Participants) | 121
  7-years Mental Component: number analyzed (hips) | 130
  7-years Mental Component | 55.53 (7.94)
  10-years Mental Component: number analyzed (Participants) | 51
  10-years Mental Component: number analyzed (hips) | 54
  10-years Mental Component | 55.73 (8.4)

8. Secondary Outcome: Lower Extremity Activity Scale (LEAS) Improvement From Preoperative Score
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: preop, 6 week, 1,2,3,4,5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
score on a scale
  Pre-op | 9.2 (3.06)
  6 weeks: number analyzed (Participants) | 322
  6 weeks: number analyzed (hips) | 340
  6 weeks | 8.94 (2.59)
  1-year: number analyzed (Participants) | 290
  1-year: number analyzed (hips) | 309
  1-year | 11.49 (2.94)
  2-years: number analyzed (Participants) | 259
  2-years: number analyzed (hips) | 277
  2-years | 11.79 (3.09)
  3-years: number analyzed (Participants) | 224
  3-years: number analyzed (hips) | 241
  3-years | 11.82 (2.96)
  4-years: number analyzed (Participants) | 202
  4-years: number analyzed (hips) | 218
  4-years | 11.66 (2.99)
  5-years: number analyzed (Participants) | 199
  5-years: number analyzed (hips) | 213
  5-years | 11.62 (2.99)
  7-years: number analyzed (Participants) | 123
  7-years: number analyzed (hips) | 132
  7-years | 11.3 (3.17)
  10-years: number analyzed (Participants) | 54
  10-years: number analyzed (hips) | 57
  10-years | 10.84 (3.21)

9. Secondary Outcome: EQ-5D Index Score Improvement From Preoperative Score
Description: The EQ-5D is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; the EQ visual analogue scale (EQ VAS) and EQ-5D descriptive system. The EQ VAS collects health state values using a 20 cm visual analogue scale with the endpoints labeled best imaginable health state at the top and worst imaginable health state at the bottom, having numeric values of 100 to 0 respectively. The EQ-5D Time Trade-off (TTO) descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/comfort and anxiety/depression. Each dimension has three levels: no problems, some problems and extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health, and a high score shows better health.
Time Frame: preop, 6 week, 1,2,3,4,5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
score on a scale
  EQ-5D Pre-op: number analyzed (Participants) | 213
  EQ-5D Pre-op: number analyzed (hips) | 224
  EQ-5D Pre-op | 67.22 (19.16)
  EQ-5D 6 weeks: number analyzed (Participants) | 208
  EQ-5D 6 weeks: number analyzed (hips) | 220
  EQ-5D 6 weeks | 78.58 (15.53)
  EQ-5D 1-year: number analyzed (Participants) | 236
  EQ-5D 1-year: number analyzed (hips) | 250
  EQ-5D 1-year | 82.9 (13.76)
  EQ-5D 2-years: number analyzed (Participants) | 231
  EQ-5D 2-years: number analyzed (hips) | 245
  EQ-5D 2-years | 83.89 (13.14)
  EQ-5D 3-years: number analyzed (Participants) | 209
  EQ-5D 3-years: number analyzed (hips) | 222
  EQ-5D 3-years | 84.14 (12.29)
  EQ-5D 4-years: number analyzed (Participants) | 186
  EQ-5D 4-years: number analyzed (hips) | 200
  EQ-5D 4-years | 83.18 (12.54)
  EQ-5D 5-years: number analyzed (Participants) | 185
  EQ-5D 5-years: number analyzed (hips) | 198
  EQ-5D 5-years | 81.26 (14.63)
  EQ-5D 7-years: number analyzed (Participants) | 120
  EQ-5D 7-years: number analyzed (hips) | 128
  EQ-5D 7-years | 80.5 (16.21)
  EQ-5D 10-years: number analyzed (Participants) | 48
  EQ-5D 10-years: number analyzed (hips) | 50
  EQ-5D 10-years | 81.58 (21.09)
  E-5D TTO Pre-op: number analyzed (Participants) | 213
  E-5D TTO Pre-op: number analyzed (hips) | 224
  E-5D TTO Pre-op | 0.63 (0.19)
  EQ-5D TTO 6 weeks: number analyzed (Participants) | 208
  EQ-5D TTO 6 weeks: number analyzed (hips) | 220
  EQ-5D TTO 6 weeks | 0.81 (0.15)
  EQ-5D TTO 1-year: number analyzed (Participants) | 236
  EQ-5D TTO 1-year: number analyzed (hips) | 250
  EQ-5D TTO 1-year | 0.89 (0.13)
  EQ-5D TTO 2-years: number analyzed (Participants) | 233
  EQ-5D TTO 2-years: number analyzed (hips) | 247
  EQ-5D TTO 2-years | 0.90 (0.13)
  EQ-5D TTO 3-years: number analyzed (Participants) | 208
  EQ-5D TTO 3-years: number analyzed (hips) | 221
  EQ-5D TTO 3-years | 0.91 (0.13)
  EQ-5D TTO 4-years: number analyzed (Participants) | 193
  EQ-5D TTO 4-years: number analyzed (hips) | 208
  EQ-5D TTO 4-years | 0.9 (0.13)
  EQ-5D TTO 5-years: number analyzed (Participants) | 187
  EQ-5D TTO 5-years: number analyzed (hips) | 200
  EQ-5D TTO 5-years | 0.89 (0.15)
  EQ-5D TTO 7-years: number analyzed (Participants) | 120
  EQ-5D TTO 7-years: number analyzed (hips) | 128
  EQ-5D TTO 7-years | 0.9 (0.13)
  EQ-5D TTO 10-years: number analyzed (Participants) | 49
  EQ-5D TTO 10-years: number analyzed (hips) | 51
  EQ-5D TTO 10-years | 0.92 (0.17)

10. Secondary Outcome: Percentage of Cases Which Did Not Have Any Component Revised
Description: The number of hips that did not undergo a removal/revision of any of the hip components.
Time Frame: 10 years
Population: Participants/hips with available data at 10 years or at the time of early study termination. There were 12 hip revisions of the 354 hips in the study, leaving 342 hip cases without a revision of any components.
Measure: Number; unit: hips
Units Other Than Participants: hips
Arm/Group | Restoration ADM X3 Device
Number analyzed (Participants) | 333
Number analyzed (hips) | 354
hips | 342

ADVERSE EVENTS:
Time Frame: The study period during which AEs must be reported is defined as the period from the initiation of any study procedures to the end of the study treatment follow-up. The start of study procedures is considered to be the date of consent. Any AEs that meet the protocol defined reportable events must be reported from the time of consent through study completion (10 years) or in this case early study termination.
Description: Serious systemic adverse events (excluding elective procedures), and all AEs, whether serious or not, related to the operative site were collected. Date of occurrence, date diagnosed, type of complication and treatment was collected. Industry standard AE and SAE terms were used in the study.
Groups:
- Operative Site Events: All adverse events whether serious or not that occurred within the study population of 354 hips. These events are reported by unit/hip because in the case of bilateral participants (when one participant has both hips enrolled in the study), an event can occur in one hip, both hips or the same hip at different times and are counted separately (by hip) for this reason.
- Non Operative Site Events: All serious systemic adverse events that occurred in the study population of 333 participants.
Arm/Group | Operative Site Events | Non Operative Site Events
All-Cause Mortality (participants affected / at risk) | 0/354 | 13/333
Serious Adverse Events (participants affected / at risk) | 15/354 | 66/333
Other Adverse Events (participants affected / at risk) | 56/354 | 0/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Site Events (N=354) | Non Operative Site Events (N=333)
Non-operative site (Blood and lymphatic system disorders) | 0/0 (0) | 4 (4) — Anemia, Leukemia
Non-operative site (Cardiac disorders) | 0/0 (0) | 9 (13) — Bradycardia, Aortic Stenosis, Syncopal Episode, Stemi, Atrial Flutter, Embolism of Left Middle Cerebral Artery, A-fib, Quadruple Bypass Surgery, Paroxysmal Atrial Fibrillation, Tachycardia
Non-operative site (Endocrine disorders) | 0/0 (0) | 1 (1) — Hypothyroidism
Non-operative site (Gastrointestinal disorders) | 0/0 (0) | 9 (9) — Cholecystectomy, Inguinal Hernia, Hiatal Hernia, Bowel Obstruction, Ruptured Intestine
Non-operative site (Hepatobiliary disorders) | 0/0 (0) | 1 (1) — Liver Cirrhosis
Non-operative site (Infections and infestations) | 0/0 (0) | 7 (8) — Sepsis, Abscess, Bacteremia, Pneumonia, Acute COPD Bronchitis
Non-operative site (Injury, poisoning and procedural complications) | 0/0 (0) | 4 (5) — Thoracic Spine Compression Fracture, Wound Hematoma
Operative site (Injury, poisoning and procedural complications) | 3 (3) | 0/0 (0) — Fall Operative Side, Soft Tissue Trauma, Hip Fracture
Non-operative site (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1) — Hypernatremia
Operative site (Musculoskeletal and connective tissue disorders) | 11 (14) | 0/0 (0) — Femur Fracture, Hip Pain, Trochanteric Bursitis, Tibial Plateau Fracture, Soft Tissue Trauma, Tendonitis, Muscle Repair, Femoral Component Loosening, Metallosis
Non-operative site (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 12 (12) — Shoulder Impingement, Thoracic Spine Fracture, Spinal Stenosis, Spinal Fusion,
Non-operative site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 13 (13) — Lung Cancer, Myeloblastoma of the brain, Pancreatic cancer, Prostate cancer, Renal Cancer, Breast Cancer
Operative site (Nervous system disorders) | 1 (1) | 0/0 (0) — Nerve Palsy
Non-operative site (Nervous system disorders) | 0/0 (0) | 2 (2) — Alzheimer's Dementia, Acute Intracerebral Hemorrhage
Non-operative site (Renal and urinary disorders) | 0/0 (0) | 4 (4) — UTI, Chronic Renal Insufficiency, Worsening Renal Function, Kidney Cancer
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 4 (4) — Lung Cancer, Pneumonia, Pulmonary Embolism, Difficulty Breathing
Non-operative site (Surgical and medical procedures) | 0/0 (0) | 2 (2) — Ulcus Left Thorax, Trauma
Non-operative site (Vascular disorders) | 0/0 (0) | 7 (7) — DVT, Stroke, Atherosclerosis, Pulmonary Embolism, Coronary Artery Disease
Non-operative site (General disorders) | 0/0 (0) | 6 (6) — Generalized weakness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Site Events (N=354) | Non Operative Site Events (N=333)
Operative site (Musculoskeletal and connective tissue disorders) | 56 (62) | 0/0 (0)

LIMITATIONS AND CAVEATS:
Due to circumstances starting with the COVID-19 pandemic and challenges recalling study subjects for long term postoperative visits, the follow-up compliance decreased significantly. Therefore, there would be inadequate subjects to analyze at the 10 year endpoint. For this reason, a business decision was made to close the study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each study investigator has independent publication privileges for their own center's results after multi-center publications are submitted. Sponsor requires review of publications. Sponsor shall not edit or influence the publications except to ensure that confidential information is not disclosed, no off-label device use is promoted, and that data is accurately represented. Any publications must be submitted to Stryker for review at least 60 days prior to submission of publication.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT01420237/Prot_SAP_ICF_000.pdf